CLINICAL TRIAL: NCT07191223
Title: Evaluation of Knowledge on Tick-borne Encephalitis Virus (TBEV) Infection Among General Practitioners and Specialists in Endemic Areas and Outside Endemic Areas in France
Brief Title: Evaluation of Knowledge on Tick-borne Encephalitis Virus (TBEV) Infection Among General Practitioners in France
Acronym: CoMTBEV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9141
Record Dates: First submitted 2025-03-25; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: Tick-borne Encephalitis, France
Keywords: Tick-borne encephalitis; tick bite
MeSH Terms: conditions — Encephalitis, Tick-Borne; Tick Bites

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tick-borne encephalitis is a relatively rare disease (approximately 35 cases diagnosed per year), but most cases (86%) are due to contamination in France via a tick bite. Of the 71 cases reported over two years (May 2021 to May 2023), 94% of patients were hospitalized.

It is therefore important to consider and diagnose at the first signs to ensure appropriate follow-up and also to implement primary prevention in endemic/at-risk areas.

ELIGIBILITY:
Inclusion Criteria:

* Be a doctoral student or in training
* Practice in France
* Agree to participate in the survey.

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Doctoral student or in training and practicing in France
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
Tick-borne meningoencephalitis knowledge score | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Service des maladies infectieuses et tropicales - CHU de Strasbourg - France, Strasbourg, France